CLINICAL TRIAL: NCT07330596
Title: A Randomized Controlled Study Comparing the Efficacy of QL1706 Combined With Chemotherapy in the Treatment of Immune-mediated Non-small Cell Lung Cancer
Brief Title: QL1706 Combined With Chemotherapy in the Treatment of Immune-mediated NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Provincial Cancer Hospital (Other)
Responsible Party: Principal Investigator, Shuanghu Yuan, Professor, Anhui Provincial Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRAD2
Record Dates: First submitted 2025-06-27; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: NSCLC (Advanced Non-small Cell Lung Cancer)
Keywords: NSCLC; Immune resistance; PD-1/CTLA-4; EGFR/ALK Mutation Negative
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: This study is a prospective, multicenter, open label randomized controlled trial design, recruiting 96 immunocompromised driver gene negative patients with locally advanced or recurrent/metastatic non-small cell lung cancer. The experimental group received QL1706 combined with docetaxel or gemcitabine treatment in a 1:1 ratio, while the control group received docetaxel or gemcitabine treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- QL1706 combined with chemotherapy (Experimental): QL1706：5mg/kg，iv，d1 combined with Gemcitabine (1000mg/m2，iv，d1、d8 )or DOCETAXEL (60mg/m2，iv，d1)
  Interventions: Drug: QL1706 combined with Chemotherapy
- chemotherapy (Active Comparator): Gemcitabine (1000mg/m2，iv，d1、d8 )or DOCETAXEL (60mg/m2，iv，d1)
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: QL1706 combined with Chemotherapy — QL1706：5mg/kg，iv，d1 combined with Gemcitabine (1000mg/m2，iv，d1、d8 )or DOCETAXEL (60mg/m2，iv，d1)
  Arms: QL1706 combined with chemotherapy
Drug: Chemotherapy — Gemcitabine (1000mg/m2，iv，d1、d8 )or DOCETAXEL (60mg/m2，iv，d1)
  Arms: chemotherapy

SUMMARY:
Lung cancer is the leading cause of cancer-related deaths worldwide. According to the 2023 global cancer statistics, there are approximately 2.47 million new cases and 1.76 million deaths of lung cancer annually, accounting for 18.4% of all cancer deaths. Among them, driver gene negative NSCLC accounts for about 30% -40% of all NSCLC. In China, the incidence rate and mortality of lung cancer rank first. In 2022, there will be about 870000 new cases and 760000 deaths. In Chinese NSCLC patients, the EGFR mutation rate is about 50%, ALK fusion is about 5%, other mutations (ROS1, RET, etc.) are about 5% -10%, and the negative proportion of driver genes is about 30% -40%. Traditional treatment for late stage non-small cell lung cancer with negative driver genes has limited clinical efficacy. In recent years, the emergence of immune checkpoint inhibitors (ICIs) has greatly changed the treatment pattern of advanced non-small cell lung cancer patients, significantly prolonging the overall survival of advanced cancer patients. For the follow-up treatment of patients with previous immunotherapy, the current standard treatment regimen is still mainly chemotherapy. However, these plans have mediocre efficacy and significant side effects, making it difficult to meet the current clinical treatment needs. At present, there is no unified treatment plan for first-line immunotherapy or immunotherapy combined with chemotherapy in patients with driver gene negative advanced NSCLC. Second line chemotherapy such as docetaxel is currently recommended as the standard treatment plan in NCCN guidelines and CSCO guidelines. Research suggests that for patients with first-line immune resistance or immune combined chemotherapy resistance, second-line immune re challenge can still bring certain survival benefits to patients, but the benefits are limited and new treatment options need to be explored.

Iparomlimab injection (drug number QL-1706) is a novel combination antibody independently developed by Qilu Company. It consists of Iparomlimab, an IgG4 antibody targeting PD-1, and Tuvonralimab, an IgG1 antibody targeting CTLA-4, in a fixed ratio. It has a synergistic mechanism of simultaneously blocking PD-1 and CTLA-4. In summary, ICIs are still an important treatment strategy for advanced non-small cell lung cancer. However, the emergence of drug resistance after immunotherapy seriously affects the survival time and prognosis of patients. Preliminary research has been conducted on the resistance mechanism of immunotherapy, but more research is needed to clarify the main mechanisms of action, in order to further prevent and overcome drug resistance. QL1706 has shown promising preliminary efficacy and good tolerability in PD-1 resistant NSCLC in preclinical and phase I clinical studies. Based on this, this study aims to conduct an exploratory study on QL1706 combined with chemotherapy compared to chemotherapy alone in the treatment of immune regulated non-small cell lung cancer with negative driver genes.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, open label randomized controlled trial design, recruiting 96 immunocompromised driver gene negative patients with locally advanced or recurrent/metastatic non-small cell lung cancer. The experimental group received QL1706 combined with docetaxel or gemcitabine treatment in a 1:1 ratio, while the control group received docetaxel or gemcitabine treatment.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in the research and sign an informed consent form; Age ≥ 18 years old, ≤ 75 years old;
* Diagnosed with NSCLC through histology or cytology;
* No EGFR sensitive mutations or ALK gene translocation changes;
* Previously received PD-1/PD-L1 inhibitors combined with platinum based dual therapy or sequential therapy as first-line treatment for advanced metastatic or recurrent NSCLC, and disease progression occurred during or after treatment; At least one measurable lesion should be used as the target lesion (RECIST v1.1 standard);
* ECOG score: 0-2 points;
* Expected survival period is not less than 12 weeks;
* Women of childbearing age must undergo a pregnancy test (serum or urine) with a negative result within 28 days before enrollment, and voluntarily use appropriate contraception methods during the observation period and within 8 weeks after the last dose; For males, surgical sterilization or consent to use appropriate contraception methods during the observation period and within 8 weeks after the last dose should be provided;
* The laboratory test results during the screening period indicate that the patient has good organ function: a) Hematology (no blood transfusion within 14 days and no treatment with blood components or granulocyte colony-factor): Neutrophil count (NEU) ≥ 1.5 × 10 ^ 9/L (1500/mm3); Platelet count (PLT) ≥ 100 × 10 ^ 9/L (100000/mm3); Hemoglobin ≥ 90 g/L; b) Liver: serum total bilirubin (TBil) ≤ ULN; Glutamate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 1.5 × ULN; AST or ALT should be 1.5-3.5 × ULN, and alkaline phosphatase (ALP) should be ≤ 2.5 × ULN; c) Kidney: creatinine clearance rate (CrCl) calculated value ≥ 30 mL/min; d) Coagulation function: International normalized ratio (INR) ≤ 1.5, and prothrombin time (PT) or activated partial thromboplastin time (APTT) ≤ 1.5 × ULN; j) International Normalized Ratio (INR) ≤ 1.5; Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN;
* Patients whom researchers believe can benefit.

Exclusion Criteria:

* There are EGFR sensitive mutations or ALK gene translocation changes present;
* Previously received PD1/CTLA4 bispecific antibody therapy;
* Adverse reactions caused by previous treatment have not recovered to CTCAE (version 5.0) grade 1 or below (excluding toxicity ≤ grade 2 that has been determined by the researcher to exist for a long time, cannot be recovered, and does not increase safety risks);
* Symptomatic central nervous system metastasis. Patients who have received treatment for brain metastases and have been deemed stable by researchers may consider participating in this study;
* For patients with poor control of cancer-related pain, those who require analgesic treatment must receive a stable dose of treatment before participating in the study;
* Chest fluid, ascites or pericardial effusion with clinical symptoms or unstable condition after symptomatic treatment;
* Known to have a history of severe allergic reactions to the drug and its components, planned chemotherapy drugs, and those with a history of severe allergic reactions;
* Suffering from or suspected of active autoimmune diseases, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory intestinal diseases, etc., except: type I diabetes and hypothyroidism that can be controlled through stable dose replacement treatment, and skin diseases that do not require systemic treatment (such as psoriasis, vitiligo);
* History of interstitial lung disease or drug-induced interstitial lung disease or pneumonia in the past;
* Corticosteroid drugs (prednisone>10mg/day or equivalent dose) or other immunosuppressive drugs received systemically within 14 days prior to the first study medication;
* Individuals with a history of immunodeficiency, including those with other acquired or congenital immunodeficiency diseases, those with a history of organ transplantation, or those who have received allogeneic hematopoietic stem cell transplantation or solid organ transplantation; Received live vaccination within 4 weeks before the first study medication;
* Suffering from serious cardiovascular and cerebrovascular diseases: a) poorly controlled hypertension or pulmonary arterial hypertension; b) Unstable angina or myocardial infarction, coronary artery bypass grafting or stent implantation within 6 months prior to study medication; c) Chronic heart failure with heart function ≥ 2 (NYHA classification by the New York Heart Association); d) Left ventricular ejection fraction (LVEF)<50%; e) Various severe arrhythmias requiring medication treatment (excluding atrial fibrillation or paroxysmal supraventricular tachycardia). For example, male QTcF>450 milliseconds or female QTcF>470 milliseconds, complete left bundle branch block, grade III block; f) Cerebrovascular accident (CVA) or transient ischemic attack (TIA) occurred within 6 months prior to the study medication;
* Positive result of human immunodeficiency virus (HIV) antibody test, active hepatitis B or C. The following conditions are allowed to participate in this study: a) hepatitis B core antibody (HBcAb) or hepatitis B surface antigen (HBsAg) is positive, but HBV DNA is lower than the lower limit of the detection value of the research center (negative) or less than 500IU/ML, and the active infection is excluded according to the judgment of the researcher based on clinical treatment and performance; b) Individuals with positive hepatitis C antibodies and HCV RNA below the lower limit (negative) of the detection value at the research center;
* Suffering from other active malignant tumors other than the research disease within 5 years, except for malignant tumors that can be expected to recover after treatment (including but not limited to fully treated thyroid cancer, cervical carcinoma in situ, basal or squamous cell carcinoma, or breast ductal carcinoma in situ treated with radical surgery);
* Individuals with a history of substance abuse and inability to quit, or those with a history of mental disorders;
* Pregnant or lactating women;
* The researcher believes that the patient is not suitable to participate in any other circumstances of this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2028-01-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
PFS | "From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months"
  Refers to the time from the start of medication to the first occurrence of disease progression or death from any cause

SECONDARY OUTCOMES:
ORR | through study completion, an average of 1 year
  It refers to the proportion of patients whose tumor volume shrinks by 30% and can be maintained for more than four weeks, that is, the proportion of subjects who achieve complete response (CR) and partial response (PR)
DCR | through study completion, an average of 1 year
  It refers to the proportion of subjects who achieve complete remission (CR), partial remission (PR), and disease stability (SD) at the end of treatment
DOR | through study completion, an average of 1 year
  Refers to the time from the first judgment of complete remission (CR) or partial remission (PR) to the discovery of disease progression (PD)
OS | through study completion, an average of 1 year
  It refers to the time from the start of medication to death caused by any reason
AE | through study completion, an average of 1 year
  AE

CONTACTS AND LOCATIONS:
Overall Officials: shuanghu yuan, MD, Study Chair — Anhui Provincial Cancer Hospital
Locations (1):
- Anhui cancer hospital, Hefei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Franchi M, Pellegrini G, Corrao G. Effectiveness and Cost-Effectiveness Profile of Second-Line Treatments with Nivolumab, Pembrolizumab and Atezolizumab in Patients with Advanced Non-Small Cell Lung Cancer. Pharmaceuticals (Basel). 2022 Apr 18;15(4):489. doi: 10.3390/ph15040489. PMID 35455486
- [Result] 19. Hellmann MD, et al. Nivolumab plus Ipilimumab in NSCLC. NEJM. 2019.
- [Result] 18. Wang J, et al. Phase I Trial of QL1706 in Solid Tumors. ASCO. 2023 (Abstract 2505).
- [Result] 17. Wang J, et al. QL1706 + Chemotherapy in PD-1 Resistant NSCLC Models. AACR Annual Meeting. 2023 (Abstract LB002).
- [Result] DOI:https://doi.org/10.1016/j.annonc.2022.07.1146.
- [Result] Reckamp KL, Redman MW, Dragnev KH, Minichiello K, Villaruz LC, Faller B, Al Baghdadi T, Hines S, Everhart L, Highleyman L, Papadimitrakopoulou V, Neal JW, Waqar SN, Patel JD, Gray JE, Gandara DR, Kelly K, Herbst RS. Phase II Randomized Study of Ramucirumab and Pembrolizumab Versus Standard of Care in Advanced Non-Small-Cell Lung Cancer Previously Treated With Immunotherapy-Lung-MAP S1800A. J Clin Oncol. 2022 Jul 20;40(21):2295-2306. doi: 10.1200/JCO.22.00912. Epub 2022 Jun 3. PMID 35658002
- [Result] DOI: 10.1200/JCO.2021.39.15_suppl.9073.
- [Result] From the American Association of Neurological Surgeons (AANS), American Society of Neuroradiology (ASNR), Cardiovascular and Interventional Radiology Society of Europe (CIRSE), Canadian Interventional Radiology Association (CIRA), Congress of Neurological Surgeons (CNS), European Society of Minimally Invasive Neurological Therapy (ESMINT), European Society of Neuroradiology (ESNR), European Stroke Organization (ESO), Society for Cardiovascular Angiography and Interventions (SCAI), Society of Interventional Radiology (SIR), Society of NeuroInterventional Surgery (SNIS), and World Stroke Organization (WSO); Sacks D, Baxter B, Campbell BCV, Carpenter JS, Cognard C, Dippel D, Eesa M, Fischer U, Hausegger K, Hirsch JA, Shazam Hussain M, Jansen O, Jayaraman MV, Khalessi AA, Kluck BW, Lavine S, Meyers PM, Ramee S, Rufenacht DA, Schirmer CM, Vorwerk D. Multisociety Consensus Quality Improvement Revised Consensus Statement for Endovascular Therapy of Acute Ischemic Stroke. Int J Stroke. 2018 Aug;13(6):612-632. doi: 10.1177/1747493018778713. Epub 2018 May 22. No abstract available. PMID 29786478
- [Result] DOI: https://doi.org/10.1016/j.jtho.2022.07.043.
- [Result] Park SE, Lee SH, Ahn JS, Ahn MJ, Park K, Sun JM. Increased Response Rates to Salvage Chemotherapy Administered after PD-1/PD-L1 Inhibitors in Patients with Non-Small Cell Lung Cancer. J Thorac Oncol. 2018 Jan;13(1):106-111. doi: 10.1016/j.jtho.2017.10.011. Epub 2017 Oct 31. PMID 29101058
- [Result] Diker O, Olgun P. Salvage chemotherapy in patients with nonsmall cell lung cancer after prior immunotherapy: a retrospective, real-life experience study. Anticancer Drugs. 2022 Sep 1;33(8):752-757. doi: 10.1097/CAD.0000000000001330. Epub 2022 Aug 10. PMID 35946540
- [Result] Muto S, Inomata S, Yamaguchi H, Mine H, Takagi H, Watanabe M, Ozaki Y, Inoue T, Yamaura T, Fukuhara M, Okabe N, Matsumura Y, Hasegawa T, Osugi J, Hoshino M, Higuchi M, Shio Y, Suzuki H. [Resistance Mechanisms to Immune Checkpoint Inhibitor and Its Overcome with Focus on beta-Catenin in Lung Cancer]. Gan To Kagaku Ryoho. 2022 Sep;49(9):928-931. Japanese. PMID 36156007
- [Result] 7. DOI: 10.1200/JCO.19.00934.
- [Result] Dafni U, Tsourti Z, Vervita K, Peters S. Immune checkpoint inhibitors, alone or in combination with chemotherapy, as first-line treatment for advanced non-small cell lung cancer. A systematic review and network meta-analysis. Lung Cancer. 2019 Aug;134:127-140. doi: 10.1016/j.lungcan.2019.05.029. Epub 2019 May 30. PMID 31319971
- [Result] Huang MY, Jiang XM, Wang BL, Sun Y, Lu JJ. Combination therapy with PD-1/PD-L1 blockade in non-small cell lung cancer: strategies and mechanisms. Pharmacol Ther. 2021 Mar;219:107694. doi: 10.1016/j.pharmthera.2020.107694. Epub 2020 Sep 25. PMID 32980443
- [Result] 3. Wu YL, et al. Genomic Landscape of Chinese Lung Cancer Patients. J Thorac Oncol. 2020.
- [Result] 2. Zheng RS, et al. Cancer Incidence and Mortality in China, 2022. JNCC. 2023
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338

DOCUMENTS (1):
  • Study Protocol (2025-04-21): https://cdn.clinicaltrials.gov/large-docs/96/NCT07330596/Prot_000.pdf